CLINICAL TRIAL: NCT02272933
Title: Operability and Implementation of a Patient Motion Monitoring System Using Wireless Body Worn Sensors
Acronym: GFD1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Study Enrollment
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: L14-125
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Accidental Falls; Gait, Unsteady
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wireless Body-Worn Sensors (Experimental): Elderly patients will wear sensors (Smart Slippers and a belt-clip sensor) as they go about their daily life in a geriatric care center.
  Interventions: Device: Smart Slipper; Device: Belt-Clip Sensor

INTERVENTIONS:
Device: Smart Slipper — The shoe measures foot pressure and motion allowing gait to be quantified.
Device: Belt-Clip Sensor — The sensor measures acceleration of the body allowing falls to be detected.

SUMMARY:
In this observational study, a motion monitoring system including body-worn sensors, communication portals, data capture system, and algorithms will be tested with geriatric patients in Garrison Geriatric Education and Care Center (Lubbock, TX). The study is part of a long-term effort to improve the quality of life and safety of geriatric patients by using autonomous systems that can alert care givers of mobility issues and falls.

DETAILED DESCRIPTION:
Medical monitoring systems have become an important area of research and development due to the possibility of allowing improved quality of life and care while reducing overall medical costs.

Significance of the study:

The study is significant because it will allow researchers to understand the efficacy of the autonomous sensor system used with actual residents of a geriatric care center. This study is one of the first attempts to monitor movements of geriatric residents as they go about their activities of daily living. This type of system has the potential to improve the quality of life and safety of geriatric patients.

Goals:

The development of autonomous patient monitoring technologies that will eventually improve the quality of life and safety of patients in geriatric care facilities and other environments.

Determine the performance and usability of the wearable sensor system in a geriatric care facility with actual residents going about their daily lives.

Specific Aims:

1. Determine performance of motion data collect ion system for monitoring geriatric residents as they go about their daily life in a geriatric center
2. Determine tolerability of wearing sensors by geriatric residents
3. Understand how medical staff interacts with monitored residents and the sensor devices
4. Determine if the sensor system's algorithms can identify falls

Objectives:

1. Analyze the motion data generated by the system to determine system performance. The list of performance metrics will include: (a) system up-time, (b) continuity of data collection (c) sensor device failure rate, (d) sensor device battery life (e) simultaneous collection of data when multiple monitored residents are in the same localized area.
2. Assess the tolerability of wearing the devices over the course of a day using a survey administered to residents.
3. Assess the usability of the sensor system using a survey administered to care givers.
4. Compare events flagged as falls by system algorithms with the fall log produced by Garrison staff, cross-verified against personal fall logs, to determine the ability of the system to detect falls.

ELIGIBILITY:
Inclusion Criteria:

1. At least 30 day resident of Garrison.
2. Deemed mentally competent by primary care provider to make decisions regarding their daily shoe wear.
3. A resident prone to falls is eligible.
4. Willing to wear shoes and offer high level of compliance to study
5. Able to provide informed consent
6. Able to complete survey
7. Age range: 45-85 yrs

Exclusion Criteria:

1. Unwilling to participate 2. Not mentally competent to provide informed consent

-

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Detection of Fall Incidences | 6 months
  Participants will be monitored for falls. The detection of fall events as determined by the sensors will be compared to the fall log kept by Garrison Geriatric Center.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Banister, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Garrison Geriatric Education and Care Center, Lubbock, Texas, United States